CLINICAL TRIAL: NCT03987165
Title: The Effect of Music Therapy on Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1043190
Record Dates: First submitted 2019-06-06; First posted 2019-06-14 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Neonatal Abstinence Syndrome; Substance Withdrawal, Neonatal
Keywords: Neonatal Opioid Withdrawal Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: cross over design with each baby serving as its own control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): Music therapy by a certified music therapist will be delivered to infants over a period of 5 days. There will be two periods of data collection each day, one in the morning and one in the afternoon. Each baby will receive music therapy during one of these time points, with each baby serving as their own control during the second timepoint.
  Interventions: Other: Music Therapy
- Control (No Intervention)

INTERVENTIONS:
Other: Music Therapy — Music therapy will be conducted once daily using a Song of Kin, a familiar song used to lull the infant to sleep. If no Song of Kin is provided, "Twinkle Twinkle Little Star" will be the default lullaby.
  Arms: Music Therapy

SUMMARY:
The clinical study is evaluating the impact of music therapy on neonates, specifically infants with neonatal opioid withdrawal syndrome (NOWS). The goal is to study the effect of music therapy on an infant's behavioral (i.e feeding patterns, sleep patterns, severity of withdrawal) and physiological systems (i.e. heart rate, respiratory rate). The investigators are also studying the impact of music therapy on the infant's utilization of resources (i.e. total opioid usage and total length of stay).

DETAILED DESCRIPTION:
The research will be carried out at the Tulane Lakeside Hospital for Women and Children. Caregivers of eligible infants will be approached by the medical team during the infants stay at the hospital and asked if they would be willing to hear more about this study. Fliers will be provided and also posted so that pregnant mothers or mothers who see the flier can also find out more about the study and decide to participate. Mothers may contact the study directly. Alternatively the medical team will ask the caregiver if the research team can contact them to set up a time to talk to them about the study. If the caregiver agrees then the contact information for the caregiver will be provided to the research team who will schedule an in person meeting to go over the protocol and obtain consent. The PI or one of the research team will meet with the infant's parent/legal guardian, review the study explaining all music therapy methods that will be used, explain the risks and benefits of participation, answer all questions and ask for consent to allow infant to participate in the study, to allow researchers to audio-video record the music therapy session, and to allow researchers to review medical records of the parent/legal guardian and infant to obtain information for the Data Collection Form regarding the infant's gestational age, race, ethnicity, gender, diagnosis, pregnancy and delivery complications, results of the any laboratory work, infant medication history, and daily withdrawal Scores over the study period, or until infant's medical discharge. Infants will still be able to participate in the study if the caregiver does not consent to audio-visual recording. Informed consent and HIPAA forms will be obtained electronically via REDCap, including electronic capture of the mother's signature as well as consenting research assistant's signature, and the original electronic copy of the informed consent and HIPAA forms are maintained in the REDCap database, accessible only by study personnel as listed in the IRB.

After informed consent has been obtained, the parent/legal guardian will complete the following questionnaires and surveys: Adverse Childhood Experiences Scale (ACE), Duke Functional Support System Questionnaire (FSSQ), Edinburgh Depression Scale (EDS), Postpartum Bonding Questionnaire (PBQ), Prenatal Life Events Scale (PLES Revised), Perinatal Stress Scale:NICU (PSS:NICU), the Coronavirus Anxiety Scale (CAS) and the COVID-19 Exposure and Family Impact Survey (CEFIS). The parent/legal guardian does not have to be present, but can be present for all music sessions.

Music therapy interventions will take place over the course of five days. The anticipated length of stay in the hospital for infants with NOWS or iatrogenic exposure to opioids is 21 days and for healthy full term infants is two to three days; however per institutional protocol, infants exposed to long-acting opioids in utero could be monitored up to 72-96 hours prior to discharge to monitor for signs of withdrawal. We will continue study procedures until completion of the music therapy treatment schedule, or until infant's discharge from the hospital if infant is discharged before completing all music therapy sessions. We will not interfere with standard medical care and therefore recognize that infants without NOWS will receive less days of music therapy in general, however the consistent daily administration of music therapy will provide some ability.

This study will use a cross-over design with participants undergoing music therapy once daily (either morning or afternoon) using a Song of Kin, defined as a familiar song used to lull the infant to sleep. If Song of Kin is not provided, the default lullaby will be "Twinkle Twinkle Little Star." In addition, there will be sessions of standard nursing care with no treatment intervention (CON). Counterbalancing will be achieved by assigning a different order of presentation of conditions for each group. Each day, infants will receive a music therapy session lasting up to 20 minutes using the above mentioned technique. The music therapy session will be in the morning or afternoon depending upon which treatment group the participant is assigned to. There will not be any visits by the music therapist during sessions that the infant is to receive standard nursing care with no treatment intervention (morning/afternoon). Over the 5 day period (all week, including weekends) participants will experience conditions in the following order (with music therapy sessions designated as "MT" and control data only designated as "C"):

Condition A:

Day 1 (AM - music therapy, PM - control) Day 2 (AM - control, PM - music therapy) Day 3 (AM - music therapy, PM - control) Day 4 (AM - control, PM - music therapy) Day 5 (AM - music therapy, PM - control)

Condition B:

Day 1 (AM - control, PM - music therapy) Day 2 (AM - music therapy, PM - control) Day 3 (AM - control, PM - music therapy) Day 4 (AM - music therapy, PM - control) Day 5 (AM - control, PM - music therapy)

Prior to the first session, a research assistant will place electrodes on the infant so that they study team can gather sympathetic and parasympathetic response non-invasively using MindWare Portable Lab System (MindWare Technologies, Gahanna, Ohio). These electrodes will remain on the infant throughout each session and be removed via adhesive removing pads following each session's data collection. This will minimize discomfort to the infant secondary to electrode removal and minimize risk of skin irritation by leaving electrodes in place for a proloned period of time. The medical team will complete the standard hospital withdrawal scoring scale for each infant with NOWS or suspected to have NOWS following unit policy. Withdrawal scores will not be collected on newborns who are not thought to have NOWS. Data related to the NOWS symptoms and medical conditions will be obtained from medical records. Additional observational data before and after the music sessions will be collected by the research assistant, including descriptions of where the session is conducted (isolette/bassinette), activity level, vital signs, sleep/wake pattern, sucking pattern, and any other observed behaviors throughout the session.

The following research materials and data collection tools are submitted with this IRB package: Data Collection Form and Key, Medical Abstraction Form, Music Therapy Session Notes, Support System Questionnaire (FSSQ), Edinburgh Depression Scale (EDS), Postpartum Bonding Questionnaire (PBQ), Prenatal Life Events Scale (PLES Revised), Adverse Childhood Experiences (ACE) Scale, Duke Functional Support System Questionnaire (FSSQ), Perinatal Stress Scale:NICU (PSS:NICU), the Coronavirus Anxiety Scale (CAS) and the COVID-19 Exposure and Family Impact Survey (CEFIS) and Research Code Identification Sheet.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the NICU or newborn nursery
2. Corrected gestational age 34 weeks or older
3. No identified hearing disorder
4. Do not have a diagnosed developmental disability (i.e. Down Syndrome)
5. Do not have Fetal Alcohol Syndrome
6. Medically cleared to participate in the study
7. Parent or legal guardian able/willing to give consent & complete surveys.

Exclusion Criteria:

1. Corrected gestational age < 34 weeks old
2. Has an identified hearing disorder
3. Has diagnosed developmental disability (i.e. Down syndrome)
4. Has Fetal Alcohol Syndrome
5. Is not medically cleared to participate in the study
6. Parent or legal guardian unable/unwilling to give consent

Ages: 1 Minute to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate | Change in average heart rate over the 20 minute sessions (both control and music therapy)
  Infant's heart rate before, during and after music therapy and during the control session.
Change in Heart Rate Variability | Change in average heart rate variability over the 20 minute sessions (both control and music therapy)
  Infant's heart rate variability before, during and after music therapy and during the control session.
Change in Sleeping Patterns | Change in phase of sleep over the 20 minute sessions (both control and music therapy)
  Basic parameters of sleeping - Type of sleep during control and intervention periods, including but not limited to, active/alert, quiet alert, sleeping. We will monitor time from end of feeding to start of sleep.
Change in Feeding Patterns | Time from feeding to onset of sleep over the 20 minute session (both control and music therapy)
  Time between the end of feeding and the onset of sleeping, with music therapy to be conducted during feeding.
Morphine Utilization | From day of birth through day of discharge, up to 6 months
  Total cumulative dosage of morphine required during the infant's hospitalization as well as the total number of days on morphine. We will also determine the day of the maximum morphine dosage required by the infant.
Total Length of Stay | From day of birth through day of discharge, up to 6 months
  The total number of days the infant was hospitalized, from day of birth to day of discharge from the NICU

CONTACTS AND LOCATIONS:
Overall Officials: Meghan P Howell, MD, Principal Investigator — Tulane University
Locations (1):
- Tulane Lakeside Hospital - Tulane University, Metairie, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pahl A, Young L, Buus-Frank ME, Marcellus L, Soll R. Non-pharmacological care for opioid withdrawal in newborns. Cochrane Database Syst Rev. 2020 Dec 21;12(12):CD013217. doi: 10.1002/14651858.CD013217.pub2. PMID 33348423